CLINICAL TRIAL: NCT01558791
Title: A Brief Educational Intervention to Improve TBI Screening Outcomes
Brief Title: A Brief Educational Intervention to Improve Traumatic Brain Injury (TBI) Screening Outcomes
Acronym: TBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 10-221
Record Dates: First submitted 2011-08-10; First posted 2012-03-20 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: TBI
Keywords: PTSD; patient education handout
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (No Intervention): Participants will be "screened as usual". These participants will have the TBI screening as usual, without the educational intervention.
- Arm 2 (Experimental): Participants will be given the TBI handout (educational intervention) along with the usual TBI screen.
  Interventions: Other: TBI handout

INTERVENTIONS:
Other: TBI handout — The intervention is an educational handout which covers key concepts found in the empirical literature and explicated in the VA/DoD mTBI practice guideline; (1) the meaning of a positive screen, (2) symptoms may be due to another condition, (3) most people with mTBI recover.
  Arms: Arm 2

SUMMARY:
This research study is designed to learn about Veterans' understanding of mild TBI (traumatic brain injury) and the VA TBI screening process. All OEF/OIF Veterans who come to one of the study-related clinics for TBI screening will be invited to participate. An educational handout on TBI will be given to half of the participants along with their TBI screening. The other half of the participants will have the usual TBI screening without the educational handout.

Veterans enrolled in the study will be asked to answer a 5-10 minute research questionnaire. The questionnaire will ask:

* About the individual: such as gender and branch of service
* About what happened during the TBI screening: such as whether the Veteran had a chance to ask the provider any questions
* About the Veteran's understanding of mild TBI: such as whether symptoms of mild TBI are long lasting

Veterans who receive the educational handout will be asked specific questions about the handout and its information.

DETAILED DESCRIPTION:
OBJECTIVE/HYPOTHESIS: The investigators propose to develop an educational handout on mild traumatic brain injury (mTBI) and to evaluate whether this brief, educational intervention improves knowledge and understanding of TBI and the screening results. The long-term goal is to promote expectations for a positive recovery in Veterans with mTBI. The specific aim is to evaluate the effect of the intervention on Veterans' knowledge and illness perceptions regarding TBI. Hypotheses are as follows:

1. Veterans who receive the educational intervention will have improved knowledge and understanding of TBI and the meaning of a positive TBI screen compared to Veterans who undergo screening as usual.
2. Veterans who screen positive for TBI and receive the educational intervention will have less negative illness perceptions regarding TBI compared to Veterans who screen positive in the control group.

Secondary analyses are to identify clinic-level barriers and facilitators to incorporation of the educational handout into the clinical encounter.

RESEARCH PLAN: The investigators will compare 2 groups of Veterans (N = 1500), half of whom are screened as usual and half of whom receive the educational intervention. Participants will be Veterans from 4 VA post-deployment clinics in Bay Pines, FL; Hampton, VA; Providence, RI; and Tampa, FL. The recruitment portion of the study will last 24 weeks at each site. The first 12 weeks of the study, all OEF/OIF Veterans that are screened for TBI will be enrolled into the screening as usual control group. The following 12 weeks all OEF/OIF Veterans screened for TBI will be enrolled into the intervention group. The investigators anticipate enrolling 750 Veterans in each group.

METHODOLOGY: All OEF/OIF Veterans screened for TBI in the 4 identified post-deployment clinics during the study period will be eligible for inclusion in the study. The primary outcome is knowledge gained about mTBI and illness perception. All participants will be given an instrument with questions on demographics and TBI knowledge and perceptions. Participants who receive the educational handout will be asked for additional feedback. The investigators will examine the effect of the intervention on the number of correct responses to the knowledge items as well as the rates of correct answers to each individual knowledge item. Further, the investigators will examine the effect of the intervention on each of the illness perception scores.

ELIGIBILITY:
Inclusion Criteria:

* All OEF/OIF Veterans screened for TBI at the designated clinic at 1 of the 4 study sites (during the 6 months of recruitment) will be eligible.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1236 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Hamblen, PhD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (5):
- United States (5):
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Screened as Usual: Participants will be "screened as usual". These participants will have the TBI screening as usual, without the educational intervention.
- TBI Handout: Participants will be given the TBI handout (educational intervention) along with the usual TBI screen.
  TBI handout: The intervention is an educational handout which covers key concepts found in the empirical literature and explicated in the VA/DoD mTBI practice guideline; (1) the meaning of a positive screen, (2) symptoms may be due to another condition, (3) most people with mTBI recover.
Period: Overall Study
Arm/Group | Screened as Usual | TBI Handout
Started | 607 | 629
Completed | 607 | 629
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All veterans screened for TBI
Groups:
- Total: Total of all reporting groups
Arm/Group | Screened as Usual | TBI Handout | Total
Number analyzed (Participants) | 607 | 629 | 1236
Age, Customized [Number; unit: participants] — Of the total study population, 7 participants did not provide their age.
  participants
    <20 years | 0 | 1 | 1
    20-29 years | 287 | 306 | 593
    30-39 years | 152 | 158 | 310
    40-49 years | 123 | 119 | 242
    50-59 years | 39 | 38 | 77
    60+ years | 5 | 1 | 6
Sex/Gender, Customized [Number; unit: participants] — Of the total study population, 69 participants did not provide their gender.
  participants
    Female | 91 | 99 | 190
    Male | 494 | 483 | 977
Marital status [Number; unit: participants] — Of the total study population, 13 participants did not provide their marital status.
  participants
    Married | 269 | 300 | 569
    Widowed | 2 | 3 | 5
    Divorced | 117 | 114 | 231
    Separated | 42 | 44 | 86
    Never married | 171 | 161 | 332
Service Branch [Number; unit: participants] — Participants were able to select all that apply, so there is overlap for those who have served in more than one service branch and those who were in the reserves. N=1231 provided information on service era.
  participants
    Army | 346 | 335 | 681
    Navy | 463 | 477 | 940
    Marine Corps | 508 | 533 | 1041
    Air Force | 524 | 543 | 1067
    National Guard | 529 | 571 | 1100
    Reserves | 570 | 581 | 1151
    Coast Guard | 599 | 617 | 1216
Employment [Number; unit: participants] — Of the total study population, 10 participants did not provide their employment status.
  participants
    Full-time | 178 | 197 | 375
    Part-time | 37 | 27 | 64
    Retired | 69 | 58 | 127
    Student | 150 | 149 | 299
    Unemployed | 170 | 191 | 361
Service connection [Number; unit: participants] — Of the total study population, 65 participants did not provide information about service connection.
  participants
    No | 305 | 277 | 582
    Yes | 278 | 311 | 589
Reported PTSD diagnosis [Number; unit: participants] — Of the total study population, 29 participants did not provide information on PTSD diagnosis.
  participants
    No | 440 | 469 | 909
    Yes | 152 | 146 | 298

OUTCOME MEASURES:

1. Primary Outcome: mTBI Questionnaire
Description: The primary outcome is knowledge gained about mTBI and illness perception. This is evaluated by number correct out of 10 true or false questions.
Time Frame: One day- Participants complete a questionnaire within 1 day of TBI screening. There is no follow up assessment.
Population: All veterans screened who accepted the questionnaire.
Measure: Mean (Standard Deviation); unit: correct answers out of 10
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 607 | 629
correct answers out of 10 | 5.38 (2.94) | 7.52 (2.65)

2. Primary Outcome: Illness Perception - Current Symptoms
Description: Participants rate on a Likert Scale from 0-10 how much their current symptoms affect their life, with 0 being no affect, and 10 being severe.
Time Frame: One day- Participants complete a questionnaire within 1 day of TBI screening. There is no follow up assessment.
Population: All veterans who accepted questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 607 | 329
units on a scale | 6.92 (2.46) | 6.79 (2.40)

3. Primary Outcome: Illness Perception - Duration of Symptoms
Description: Participants rate on a Likert Scale from 0-10 how long they think their current symptoms will continue with 0 being a very short time and 10 being forever.
Time Frame: One day- Participants complete a questionnaire within 1 day of TBI screening. There is no follow up assessment.
Population: All veterans screened who accepted questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 607 | 629
units on a scale | 7.59 (2.55) | 7.61 (2.50)

4. Secondary Outcome: Feasibility Questionnaire
Description: A brief feasibility questionnaire will be used to evaluate provider feedback regarding administering the educational handout as part of the TBI clinical reminder.
Time Frame: One month- Providers complete a questionnaire within 1 month after data collection ends for the site.
Population: PI and project staff no longer have access to this data to report results.
Arm/Group | Screened as Usual | TBI Handout
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No